CLINICAL TRIAL: NCT03971708
Title: Investigating Systemic Effects of Lidocaine Infusion for Transversus Abdominis Plane (TAP) Block Catheter
Brief Title: Systemic Effects of Lidocaine Infusion for TAP Block Catheter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00054477
Record Dates: First submitted 2019-05-29; First posted 2019-06-03 (Actual); Last update posted 2022-05-17 (Actual); Status verified 2020-06

CONDITIONS: Nephrectomy
Keywords: Lidocaine; TAP block; nephrectomy; acute pain
MeSH Terms: conditions — Acute Pain | interventions — Lidocaine; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ropivacaine (Other): This is the control where patients will receive ropivacaine via the TAP block infusion post-operatively.
  Interventions: Drug: Ropivacaine
- Lidocaine (Active Comparator): This is the study arm where patients will receive lidocaine via the TAP block infusion post-operatively.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Local anesthetic
  Other Names: Lignocaine
  Arms: Lidocaine
Drug: Ropivacaine — Local anesthetic
  Arms: Ropivacaine

SUMMARY:
Lidocaine is a local anesthetic that is usually used for nerve blocks to sensory/motor blockade. However, lidocaine can also been given intravenously, and it has been shown that this method can be used to help alleviate chronic pain. We wish to investigate if lidocaine is infused via the transversus abdominis plane (TAP) block catheter will exert systemic effect, hence reduce opioid consumption and pain score in patients compared with using local anesthetic such as ropivacaine.

DETAILED DESCRIPTION:
Following IRB approval and written consents, patients undergoing nephrectomy were randomized into 2 groups: standard 0.2% ropivacaine infusion (control) and 0.4% lidocaine infusion for TAP catheter. The TAP catheters were placed by the surgeons under direct vision at the end of surgery before wound closure. All subjects had a general anesthetic in accordance to the discretion of the anesthesiologist in the operating room. At the end of surgery, all patients received a patient-controlled analgesia (PCA) in recovery for 48 hours. The primary outcome was the total opioid consumption at the first 27 hours post-operatively. The secondary outcomes were the total opioid consumption at 4/12/24/36/48/60 hours after the initiation of local anesthetic infusion, the numerical rating scale (NRS) at rest and on movement at 4/12/24/36/48/60 hours after the initiation of the local anesthetic infusion, the incidence of nausea and vomiting, and adverse effects.

The sample size calculation for this non-inferiority trial is based on our previous retrospective study on TAP in nephrectomy patients. A sample of 80 patients is needed, using a power of 90% with the two-sided significance level of 5%. All parametric data will be analyzed using mean and standard deviation. Non-parametric data will be analyzed using median and interquartile range. Student's t-test or Mann-Whitney U test will be used to compare between groups.

ELIGIBILITY:
Inclusion Criteria:

* Elective nephrectomy
* patients consent to study
* ASA I to III

Exclusion Criteria:

* Patient refusal
* Allergy to lidocaine,
* Patients with cardiac arrhythmias or on anti-arrhythmics or propranolol
* Wolf-Parkinson White syndrome
* Hepatic disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Analgesic consumption | first 24 hours
  The amount of morphine equivalent consumption in the first 24 hours post-operatively

SECONDARY OUTCOMES:
Analgesic consumption | 4, 12, 36, 48, 72 hours
  The amount of morphine equivalent consumption 4 hours, 12 hours, 36 hours, 48 hours, and 72 hours post-operatively
Pain score | 4, 12, 24, 36, 48, 72 hours
  Pain score measured in the form of Numeric Rating Scale at 4 hours, 12 hours, 24 hours, 36 hours, 48 hours and 72 hours post-operatively

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada